CLINICAL TRIAL: NCT06042959
Title: Effects of Laughter Yoga Practiced by First Year Nursing Students Before Clinical Practice on Their Perceptions of Stress and Meaning of Life: A Randomized Controlled Trial
Brief Title: Effects of Laughter Yoga Practiced by Nursing Students Before Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MCBU-K-CEVIK-001
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy; Laughter; Stress
Keywords: Laughter therapy; Nursing; Students
MeSH Terms: conditions — Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Other: Laughter therapy

INTERVENTIONS:
Other: Laughter therapy — We used laughter yoga to investigate the potential effects on first year nursing students' whose in the preclinical period of education.
  Arms: Intervention

SUMMARY:
Aim: We conducted this randomized controlled study to determine the effect of laughter yoga practiced by first year nursing students before clinical practice on their perceptions of stress and meaning of life.

Background: Laughter yoga has a positive effect on the person's mental/general health, life satisfaction and psychological well-being and enables the person to cope with stress.

Design: In this experimental randomized and controlled study including a control group, we administered a pre-test, post-test one and post-test two to the participating students.

Methods: We conducted the study with 45 first year nursing students in the intervention group, and 45 first year nursing students in the control group. The students in the intervention group took part in eight sessions of laughter yoga for four weeks, twice a week. We used the Descriptive Information Form, Perceived Stress Scale, and Meaning and Purpose of Life Scale to collect the study data.

ELIGIBILITY:
Inclusion Criteria:

* Who did not have any diagnosed psychiatric diseases,
* Who had not done laughter yoga and / or did not have any clinical experience previously were included

Exclusion Criteria:

* Who withdrew from the study at any stage,
* Those who did not participate in the yoga sessions regularly
* Those who used another relaxation method during this period,
* Those who took antidepressants,
* Those who had a chronic cough and / or urinary incontinence,
* Those who underwent surgery in the last 3 months (abdominal surgery, uncontrolled surgery, glaucoma, hernia),
* Those who had neurological diseases such as epilepsy, multiple sclerosis,
* Those who were unwilling to participate in the study,
* Those who had neurological disorders,
* Those who lost one of their loved ones in the last 6 months were excluded from the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Meaning and Purpose of Life | four weeks
  Meaning of life of students was assessed with 17 items Meaning and Purpose of Life Scale. The options for the positive statements are scored as follows: strongly agree (5), agree (4), undecided (3), disagree (2), and strongly disagree (1). The negative statements are reverse scored. The options for the negative statements are scored as follows: strongly agree (1), agree (2), undecided (3), disagree (4) and strongly disagree (5).While the lowest possible score that can be obtained from the scale is 17, the highest possible score is 85. A high score indicates that the person's perception of the meaning and purpose of life is more positive whereas a low score indicates the person's perception of the meaning and purpose of life is more negative
Stress | four weeks
  Stress of students was assessed with Perceived Stress Scale. Responses given to the items are rated on a 5-point Likert-type scale ranging from 0 to 4 (0- Never, 1-Almost Never, 2-Sometimes, 3-Quite often, 4-Very Often). Items 4, 5, 7 and 8 containing positive statements are reverse scored. The minimum and maximum scores that can be obtained from the PSS are 0 and 40, respectively. The higher the score is the higher the level of stress is.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaya KC, Ozkan CG, Agis D. Effects of laughter yoga practiced by the first year nursing students before clinical practice on their perceptions of stress and meaning of life: a randomized controlled trial. BMC Nurs. 2025 Jan 11;24(1):41. doi: 10.1186/s12912-024-02642-0. PMID 39799345